CLINICAL TRIAL: NCT02304406
Title: RETROSPECTIVE EPIDEMIOLOGY STUDY OF ALK REARRANGEMENT IN NON-SMALL CELL LUNG CANCER PATIENTS IN THE MIDDLE EAST & NORTH AFRICA.
Acronym: ALK NSCLC MENA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081046
Record Dates: First submitted 2014-11-14; First posted 2014-12-02 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: prevalence of ALK rearrangement, NSCLC, MENA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The tissue samples of NSCLC cases will be retrieved from tissue banks of the molecular diagnostic units & pathology departments in these study centers. The histological diagnosis will be confirmed by the pathologists. The retained samples will then be tested by performing the Ventana ALK-IHC to assess the absence or presence of the ALK rearrangement by the detection of the ALK protein in formalin-fixed, paraffin-embedded NSCLC stored tissue samples using Ventana anti-ALK (D5F3) Rabbit Monoclonal Primary Antibody (Roche Diagnostics GmbH) in the selected study centers.

SUMMARY:
Thet study aims to estimate the prevalence of ALK rearrangement in the Middle East North Africa population by using the Ventana ALK-IHC method for ALK protein detection in retrospective NSCLC clinical samples, & to evaluate the association of ALK rearrangement with clinical and pathological parameters of NSCLC patients in MENA.

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional non-interventional epidemiology study to investigate the prevalence of ALK rearrangement in NSCLC patients in Middle East & North Africa. Approximately 700 retained tumor tissue specimens (tissue block) of patients previously diagnosed with NSCLC will be selected & subjected to ALK immune-staining using Ventana anti-ALK (D5F3) Rabbit Monoclonal Primary Antibody combined with OptiView Benchmark System in 6-8 centers in 5-7 countries in the MENA region.

The tissue samples of NSCLC cases will be retrieved from tissue banks of the molecular diagnostic units & pathology departments in these study centers. The histological diagnosis will be confirmed by the pathologists. The retained samples will then be tested by performing the Ventana ALK-IHC to assess the absence or presence of the ALK rearrangement by the detection of the ALK protein in formalin-fixed, paraffin-embedded NSCLC stored tissue samples using Ventana anti-ALK (D5F3) Rabbit Monoclonal Primary Antibody (Roche Diagnostics GmbH) in the selected study centers. The results of ALK testing within this study population will then be used to establish the prevalence of ALK rearrangement in MENA NSCLC patients.

The patients' characteristics, demographic, clinical and pathologic parameters will be obtained from their medical records & analyzed to determine any association with the presence of the EML4-ALK fusion gene in MENA NSCLC patients.

The assessment of concordance of the results between FISH & IHC will be done in 2-3 centers. Results of FISH testing will be collected & recorded, if the retained tissue samples had been previously tested. If not, the Vysis FISH test will be performed, to assess the concordance between the results obtained using Vysis Break-apart FISH & Ventana IHC testing methods for ALK rearrangement detection.

ELIGIBILITY:
Inclusion Criteria:

- 1. Histological confirmation of nonsquamous NSCLC, with any TNM stage. 2. Available and sufficient tissue sample for ALK testing 3.Tissue samples are less than 5 years old 4.Routinely processed formalin-fixed, paraffin-embedded tissue samples only (see exclusion criteria pertaining to tissue samples).

5.Histological sections mounted on glass slides must not be older than 3 months 6.Age > 18 years 7.Any ECOG Performance status 8.Still alive, or death confirmed before inclusion, or is unknown 9.Disease diagnosis and/or treatment in one of the centers, in the last 5 years, assigned to participate in the study; 10.Written informed consent for general investigational testing was previously obtained, or specifically obtained for this retrospective epidemiology study, or having a documented waiver for the Informed consent document use, as required by local regulatory authorities, &/or Research Ethics committee/Institutional Review Board.

Exclusion Criteria:

* 1- Tumor tissue samples older than 5 year period or samples not properly stored.

  2-Tumor tissue samples fixed by using AFA, B5, Bouin's, 95% ETOH, & alcohol fixatives.

  3-Under-fixed tissue samples (i.e. < 6 hrs) 4-Tumor tissue samples that have been subject to any decalcification processes. 5-Recycled paraffin-embedded tissue samples. 6-Cut slides stored longer than 3 months. 7-Insufficient tissue samples with less tumor cells & high amount of necrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since this is a retrospective epidemiology study, no patients will be enrolled. Tissue samples of non-squamous NSCLC cases less than 5 years old from each of the centers will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Egypt (2):
  - National Cancer Institute, Cairo
  - National Cancer Institute, Cairo / Misr Al Qadimah
- Lebanon (2):
  - American University in Beirut, Beirut
  - American University of Beirut, Beirut
- Institut National d'Oncologie, Rabat, Morocco
- Saudi Arabia (4):
  - King Abdulaziz Medical City - National Guard Hospital, Riyadh
  - King Faisal Specialty Hospital, Riyadh/Oncology Department, Riyadh
  - King Faisal Specialty Hospital, Riyadh
  - National Guard Hospital, Riyadh
- United Arab Emirates (2):
  - Tawam Hospital, Al Ain City
  - Tawam Hospital, Al Ain/Al Maqam

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081046&StudyName=Retrospective%20Epidemiology%20Study%20Of%20Eml4-alk%20Rearrangement%20In%20Non-small%20Cell%20Lung%20Cancer%20Patients%20In%20The%20Middle%20East%20%26%20North%20Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Small Cell Lung Cancer: Tissue samples of participants of Middle East North Africa (MENA) previously diagnosed with non-small cell lung cancer (NSCLC) were tested retrospectively for the prevalence of anaplastic lymphoma kinase (ALK) rearrangement.
Period: Overall Study
Arm/Group | Non-Small Cell Lung Cancer
Started | 449
Completed | 449
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: Participants above age 18 years with confirmed NSCLC, sufficient tissue sample, routinely processed formalin-fixed, paraffin-embedded)for ALK testing, with any Eastern Cooperative Oncology Group performance status, alive/death confirmed before inclusion/unknown. Diagnosed/treated in 1 of study centers.
Groups:
- Non-Small Cell Lung Cancer: Tissue samples of participants of MENA previously diagnosed with NSCLC were tested retrospectively for the prevalence of ALK rearrangement.
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 449
Age, Customized [Number; unit: Participants]
  18 to 65 years | 272
  Greater than equal to 65 years | 157
  Missing | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 308
Race/Ethnicity, Customized [Number; unit: Participants]
  Arabic | 389
  White / Caucasian | 54
  Other | 5
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prevalence of Anaplastic Lymphoma Kinase (ALK) Rearrangement
Description: Participants with prevalence of ALK rearrangement were positive for ALK: defined as presence of strong granular cytoplasmic staining in tumor cells (any percentage of positive tumor cells).
Time Frame: 3 years
Population: Full analysis set (FAS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 449
percentage of participants | 8.69 [6.26 to 11.71]

2. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Gender
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the gender of study participants.
Time Frame: 3 years
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies the participants evaluable at specific categories.
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Male: number analyzed (Participants) | 308
  Male | 10.1
  Female: number analyzed (Participants) | 140
  Female | 5.7
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.1304, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.80 to 4.77]

3. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Race
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the race of study participants.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  White /Caucasian: number analyzed (Participants) | 54
  White /Caucasian | 11.1
  Arabic: number analyzed (Participants) | 388
  Arabic | 8.5
  Others: number analyzed (Participants) | 5
  Others | 0
  Missing: number analyzed (Participants) | 1
  Missing | 0
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.6422, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Smoking History
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the smoking history of study participants as participants who never smoked, current smoker and ex-smoker.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Never: number analyzed (Participants) | 111
  Never | 9.0
  Current: number analyzed (Participants) | 133
  Current | 7.5
  Ex-smoker: number analyzed (Participants) | 86
  Ex-smoker | 5.8
  Unknown: number analyzed (Participants) | 118
  Unknown | 11.9
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.4524, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Tumor Histologic Diagnosis
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the diagnosis of tumor histology of study participants.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Adenocarcinoma: Positive: number analyzed (Participants) | 430
  Adenocarcinoma: Positive | 8.6
  Large cell carcinoma: Positive: number analyzed (Participants) | 6
  Large cell carcinoma: Positive | 16.7
  Not specified: number analyzed (Participants) | 1
  Not specified | 0
  Others: number analyzed (Participants) | 11
  Others | 9.1
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.9010, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Tumor Stage
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the tumor stage of study participants.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Stage 1: number analyzed (Participants) | 32
  Stage 1 | 6.3
  Stage 2: number analyzed (Participants) | 51
  Stage 2 | 7.8
  Stage 3: number analyzed (Participants) | 48
  Stage 3 | 6.3
  Stage 3 A: number analyzed (Participants) | 4
  Stage 3 A | 0
  Stage 3 B: number analyzed (Participants) | 10
  Stage 3 B | 10.0
  Stage 4: number analyzed (Participants) | 260
  Stage 4 | 10.0
  Missing: number analyzed (Participants) | 43
  Missing | 7.0
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.9067, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Treatment Type
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the treatment type of study participants.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Surgery with chemotherapy: number analyzed (Participants) | 53
  Surgery with chemotherapy | 7.5
  Surgery without chemotherapy: number analyzed (Participants) | 58
  Surgery without chemotherapy | 5.2
  Targeted therapy: number analyzed (Participants) | 10
  Targeted therapy | 10.0
  Chemotherapy only: number analyzed (Participants) | 154
  Chemotherapy only | 10.4
  Other: number analyzed (Participants) | 102
  Other | 7.8
  Unknown: number analyzed (Participants) | 71
  Unknown | 9.9
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.8785, Cochran-Mantel-Haenszel

8. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Progression Free Survival (PFS)
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the PFS of study participants.
Time Frame: 3 years
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 150
percentage of participants | 8.0
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.9231, Cochran-Mantel-Haenszel

9. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Line of Therapy
Description: In this outcome measure, percentage of participants with association of ALK rearrangement were evaluated and categorized in terms of the line of therapy of study participants.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  First-line: number analyzed (Participants) | 219
  First-line | 9.1
  Second-line: number analyzed (Participants) | 59
  Second-line | 8.5
  Unknown: number analyzed (Participants) | 138
  Unknown | 9.4
  Missing: number analyzed (Participants) | 32
  Missing | 3.1
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.9780, Cochran-Mantel-Haenszel

10. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Overall Response (OR)
Description: Percentage of participants with best overall response. Complete response (CR) is equal to (=) disappearance of all target lesions. Partial Response (PR) = greater than equal to (>=) 30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. Progressive disease (PD) >= 20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of the longest dimensions since treatment start, or the appearance of >= 1 new lesion. Stable disease (SD) =neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  CR: number analyzed (Participants) | 28
  CR | 14.3
  PR: number analyzed (Participants) | 15
  PR | 20.0
  PD: number analyzed (Participants) | 157
  PD | 7.6
  SD: number analyzed (Participants) | 56
  SD | 1.8
  Unknown: number analyzed (Participants) | 191
  Unknown | 9.9
  Missing: number analyzed (Participants) | 1
  Missing | 0
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.1144, Cochran-Mantel-Haenszel

11. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Participant's Status
Description: In this outcome measure participant's status at the time of sampling were evaluable for treatment-naive and treated.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Treatment-naive: number analyzed (Participants) | 415
  Treatment-naive | 8.2
  Treated: number analyzed (Participants) | 27
  Treated | 11.1
  Unknown: number analyzed (Participants) | 6
  Unknown | 33.3
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.0862, Cochran-Mantel-Haenszel

12. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Epidermal Growth Factor Receptor (EGFR) Status
Description: In this outcome measure EGFR status of participants were evaluable for not tested, wild type and mutant.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Not tested: number analyzed (Participants) | 208
  Not tested | 12.0
  Wild type: number analyzed (Participants) | 148
  Wild type | 6.8
  Mutant: number analyzed (Participants) | 61
  Mutant | 0
  Unknown: number analyzed (Participants) | 3
  Unknown | 0
  Other: number analyzed (Participants) | 28
  Other | 14.3
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.0294, Cochran-Mantel-Haenszel

13. Secondary Outcome: Percentage of Participants With Association of Anaplastic Lymphoma Kinase (ALK) Rearrangement by Knowledge Representation for Autonomous Systems (KRAS) Status
Description: In this outcome measure KRAS status of participants were evaluable for not tested, wild type, and mutant.
Time Frame: 3 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 448
percentage of participants
  Not tested: number analyzed (Participants) | 433
  Not tested | 9.0
  Wild type: number analyzed (Participants) | 6
  Wild type | 0
  Mutant: number analyzed (Participants) | 7
  Mutant | 0
  Unknown: number analyzed (Participants) | 2
  Unknown | 0
Statistical Analysis 1: Comparison: Non-Small Cell Lung Cancer; Test type: Other; p = 0.6877, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percentage Agreement Between Vysis Fluorescent In Situ Hybridization (FISH) and Ventana Immunohistochemistry (IHC) Methods for ALK Rearrangement Detection
Description: Percent overall agreement between Vysis ALK-FISH and Ventana ALK IHC tests and its 95% CI is reported in this outcome measure.
Time Frame: 3 years
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage agreement
Arm/Group | Non-Small Cell Lung Cancer
Number analyzed (Participants) | 129
percentage agreement | 98.45 [94.51 to 99.81]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events was not planned to be collected during the study
Description: Due to the non-interventional nature of the study, adverse events were not collected during the study.
Arm/Group | Non-Small Cell Lung Cancer
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT02304406/Prot_SAP_000.pdf